CLINICAL TRIAL: NCT05508087
Title: Cardiovascular Diagnostic in Assessment of Risk High Dose Chemotherapy and Hematopoietic Cell Transplantation in Patients With Haemoblasts.
Brief Title: Cardiovascular Diagnostic in Assessment of Risk HDS and HCT in Patients With Haemoblasts.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2409
Record Dates: First submitted 2022-08-15; First posted 2022-08-19 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Cardiotoxicity
Keywords: cardiotoxicity, cardiooncology, oncohematology
MeSH Terms: conditions — Cardiotoxicity | interventions — Electrocardiography; Echocardiography; Exercise Test

STUDY DESIGN:
Intervention Model Description: to evaluate the possibility of cardiovascular studies in predicting the risk of complications after autologous hematopoietic stem cell transplantation in patients with hematological malignancies
Masking Description: to evaluate the possibility of cardiovascular studies in predicting the risk of complications after autologous hematopoietic stem cell transplantation in patients with hematological malignancies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Formerly Arm Label (Other): to evaluate the possibility of cardiovascular studies in predicting the risk of complications after autologous hematopoietic stem cell transplantation in patients with hematological malignancies
  Interventions: Diagnostic Test: electrocardiography, echocardiography with the determination of global longitudinal strain, cardiopulmonary exercise test, and diagnostic of endothelial function by Angioscan

INTERVENTIONS:
Diagnostic Test: electrocardiography, echocardiography with the determination of global longitudinal strain, cardiopulmonary exercise test, and diagnostic of endothelial function by Angioscan — We use electrocardiography, echocardiography with the determination of global longitudinal strain, cardiopulmonary exercise test, and diagnostic of endothelial function by Angioscan for the prediction of cardiovascular complications after high dose chemotherapy and hematopoietic cell transplantation in patients with haemoblasts.

SUMMARY:
In this research we investigate cardiological instrumental diagnostic, such as electrocardiography, echocardiography with the determination of global longitudinal strain, cardiopulmonary exercise test, and diagnostic of endothelial function by Angioscan for the prediction of cardiovascular complications after high dose chemotherapy and hematopoietic cell transplantation in patients with haemoblasts.

DETAILED DESCRIPTION:
Cancer and cardiovascular (CV) disease are the most prevalent diseases in the developed world. Evidence increasingly shows that these conditions are interlinked through common risk factors, coincident in an ageing population, and are connected biologically through some deleterious effects of anticancer treatment on CV health. Anticancer therapies can cause a wide spectrum of short- and long-term cardiotoxic effects such as heart failure, arrhythmias, systolic and diastolic dysfunction, valvular disease, pericarditis, myocarditis, ischemic heart disease, cardiomyopathy, stroke, hypertension.

A number of studies have shown that autologous and allogeneic hematopoietic cell transplantation (HCT) contribute to an increased incidence of cardiovascular disease (CVD) and worsening of cardiovascular risk factors (CVRFs) that could contribute to further CVD over time. These observations combined with a notable increase in the number of survivors after HCT in recent years highlight the need for studies aimed at modifying risk or preventing these outcomes by changing specific approaches and/or post-HCT interventions.

The aim of this study is to evaluate the prognostic value of cardiological diagnostic, such as electrocardiography, echocardiography with the determination of global longitudinal strain, cardiopulmonary exercise test, and diagnostic of endothelial function by Angioscan for the prediction of cardiovascular complications after high dose chemotherapy and hematopoietic cell transplantation in patients with haemoblasts.

This is an observational, prospective single- centre, non-randomized study. In this research included patients with haemoblasts. Before and after hematological treatment, all patients undergo a cardiological examination, including examination, history taking, measurement of blood pressure, as well as instrumental examination, including ECG, echocardiography with the determination of global longitudinal deformation, cardiopulmonary pulmonary test, assessment of endothelial function by Angioscan. In addition, all subjects take blood for troponin T and NT-proBNP.

Patients were followed-up from 3 to 12 month after hematopoietic cell transplantation.

In this study was included patients with confirmed hemoblastosis. Written informed consent was obtained from all subjects.

Inclusion criteria were being over 18 yers of age and expected for high dose chemotherapy and hematopoietic cell transplantation, Exclusion criteria were patient's refusal.

ELIGIBILITY:
Inclusion Criteria:

* Subject being over 18 yers of age
* Subject expected for high dose chemotherapy and hematopoietic cell transplantation

Exclusion Criteria:

* Subject's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Cardiac death | Up to 5 years or in the moment of hematopoietic cell transplantation
  Cardiac death after hematopoietic cell transplantation
Death | Up to 5 years or in the moment of hematopoietic cell transplantation
  Death after hematopoietic cell transplantation

SECONDARY OUTCOMES:
All cardiovascular complications | Up to 5 years or in the moment of hematopoietic cell transplantation
  Cardiovascular complications after hematopoietic cell transplantation

OTHER OUTCOMES:
Change ejection fraction by 10% of the original | Through study completion, an average of 5 years after hematopoietic cell transplantation
  Change ejection fraction by 10% of the original after hematopoietic cell transplantation
Change GLS by 12% of the original | Through study completion, an average of 5 years after hematopoietic cell transplantation
  Change GLS by 12% of the original after hematopoietic cell transplantation
Development of diastolic dysfunction | Through study completion, an average of 5 years after hematopoietic cell transplantation
  Development of diastolic dysfunction after hematopoietic cell transplantation
Change anaerobic threshold<9,5 ml/kg/min | Through study completion, an average of 5 years after hematopoietic cell transplantation
  Change anaerobic threshold<9,5 ml/kg/min before and after hematopoietic cell transplantation
Change NTproBNP >125 mmol/l | Before and through study completion, an average of 5 years after hematopoietic cell transplantation
  Change NTproBNP >125 mmol/l before and after hematopoietic cell transplantation
Change Troponin T>14 pg/ml | Before and through study completion, an average of 5 years after hematopoietic cell transplantation
  Change Troponin T>14 pg/ml before and after hematopoietic cell transplantation
Change GLS <18% | Before hematopoietic cell transplantation
  Change GLS <18% before hematopoietic cell transplantation
Change ejection fraction <52% | Before hematopoietic cell transplantation
  Change ejection fraction <52% before hematopoietic cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Nadezhda A. Potemkina, Principal Investigator — Sechenov University
Locations (1):
- Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
According to the Local Ethics Committee's rules, we are not allowed to provide this data.